CLINICAL TRIAL: NCT00073983
Title: Phase II Study Of Sequential Gemcitabine Followed By Docetaxel For Recurrent Ewing's Sarcoma, Osteosarcoma, Or Unresectable Or Locally Recurrent Chondrosarcoma [SARC Study]
Brief Title: Gemcitabine and Docetaxel in Treating Patients With Recurrent Osteosarcoma (Closed to Accrual as of 12/21/06) or Ewing's Sarcoma or Unresectable or Locally Recurrent Chondrosarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sarcoma Alliance for Research through Collaboration (Other)
Responsible Party: Shreyaskumar Patel, MD, SARC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SARC003; NCT00070772 (obsolete NCT alias)
Record Dates: First submitted 2003-12-10; First posted 2003-12-11 (Estimated); Results first posted 2012-03-12 (Estimated); Last update posted 2012-03-12 (Estimated); Status verified 2012-02

CONDITIONS: Sarcoma
Keywords: recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; chondrosarcoma; recurrent osteosarcoma
MeSH Terms: conditions — Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Chondrosarcoma; Osteosarcoma | interventions — Filgrastim; pegfilgrastim; Docetaxel; Gemcitabine; Microarray Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: filgrastim — filgrastim
Biological: pegfilgrastim — pegfilgrastim
Drug: docetaxel — docetaxel
Drug: gemcitabine hydrochloride — gemcitabine hydrochloride
Genetic: microarray analysis — microarray analysis
Other: laboratory biomarker analysis — laboratory biomarker analysis
Other: pharmacokinetic study — pharmacokinetic study

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine and docetaxel, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining gemcitabine with docetaxel may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining gemcitabine with docetaxel in treating patients who have recurrent osteosarcoma, recurrent Ewing's sarcoma, or unresectable or locally recurrent chondrosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate in patients with recurrent osteosarcoma or Ewing's sarcoma or unresectable or locally recurrent chondrosarcoma treated with sequential gemcitabine and docetaxel.

Secondary

* Determine the time to progression in patients treated with this regimen.
* Assess the toxicity of this regimen in these patients.
* Compare the pharmacokinetics of this regimen vs gemcitabine alone in these patients.
* Obtain tumor samples for cDNA microarray analysis of gene expression and development of cell lines and xenotransplantation models.

OUTLINE: This is a nonrandomized, multicenter study.

Patients are stratified according to diagnosis recurrent osteosarcoma vs recurrent Ewing's sarcoma vs unresectable or locally recurrent chondrosarcoma).

Patients receive gemcitabine intravenously over 90 minutes on days 1 and 8 and docetaxel intravenously over 1 hour on day 8. Patients also receive filgrastim (G-CSF) subcutaneously (SC) beginning on day 9 and continuing until blood counts recover. Patients may receive pegfilgrastim SC on day 9 (once per course) as an alternative to G-CSF. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Optional blood samples are collected at baseline and periodically during study for pharmacokinetics studies. Optional tumor tissue samples from biopsy or surgical resection are analysed for cDNA microarray analysis of gene expression.

Patients are followed every 3 months for 1 year and then every 6 months for 1 year.

PROJECTED ACCRUAL: A maximum of 120 patients (40 per stratum) will be accrued for this study within 17-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed* diagnosis of 1 of the following:

  * Recurrent high-grade osteosarcoma (closed to accrual as of 12/21/06) or Ewing's sarcoma

    * Progressive disease after standard therapy
    * Received no more than 2 additional salvage regimens
  * Chondrosarcoma

    * Unresectable OR locally recurrent and unable to be completely resected NOTE: *Biopsy required for isolated pulmonary recurrences
* Measurable disease

  * At least 1 unidimensionally measurable lesion by medical imaging techniques
  * Ascites, pleural effusions, and bone marrow disease are not considered measurable disease

PATIENT CHARACTERISTICS:

Age

* 4 and over

Performance status

* ECOG (Eastern Cooperative Oncology Group) 0-2 (≥ 18 years of age)
* Karnofsky 50-100% (11-17 years of age)
* Lansky 50-100% (≤ 10 years of age)

Life expectancy

* Not specified

Hematopoietic

* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3 (transfusion independent)
* Hemoglobin ≥ 8.0 g/dL (transfusion allowed)

Hepatic

* Bilirubin ≤ upper limit of normal (ULN) (except for patients with Gilbert's syndrome)
* ALT ≤ 2.5 times ULN

Renal

* Creatinine clearance or radioisotope glomerular filtration rate > 70 mL/min/1.73 m^2 OR
* Serum creatinine ≤ ULN for age:

  * Ages 5 and under ≤ 0.8 mg/dL
  * Ages 6 to 10 ≤ 1.0 mg/dL
  * Ages 11 to 15 ≤ 1.2 mg/dL
  * Ages 16 to 18 ≤ 1.5 mg/dL

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* Sensory or motor neuropathy due to prior chemotherapy ≤ grade 1
* Sensory or motor neuropathy due to prior surgery or tumor involvement ≤ grade 2 AND stable or improving
* No active or uncontrolled infection
* No known hypersensitivity reaction to docetaxel or other polysorbate 80-formulated agents

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 72 hours since prior filgrastim (G-CSF)
* No prior allogeneic transplantation
* No concurrent immunotherapy

Chemotherapy

* At least 2 weeks since prior myelosuppressive therapy
* At least 6 months since prior myeloablative therapy
* No prior gemcitabine
* No prior taxanes
* No other concurrent chemotherapy

Endocrine therapy

* Concurrent hormonal therapy allowed

Radiotherapy

* At least 6 weeks since prior local radiotherapy
* At least 4 months since prior extensive radiotherapy to more than 50% of the pelvis
* At least 4 months since prior cranial spinal radiotherapy
* At least 6 months since prior total body irradiation
* No concurrent radiotherapy

Surgery

* No concurrent surgery

Other

* Recovered from all prior therapy
* No other concurrent investigational anticancer therapy

Min Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-10; Primary Completion 2010-01 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shreyaskumar R. Patel, MD, Principal Investigator — Sarcoma Alliance for Research through Collaboration; Elizabeth Fox, MD, Principal Investigator — Sarcoma Alliance for Research through Collaboration

REFERENCES:
- [Background] Kilgour-Christie J, Czarnecki A: Pulmonary adverse drug reactions in patients treated with gemcitabine and a combination of gemcitabine and a taxane. [Abstract] J Clin Oncol 23 (Suppl 16): A-8274, 796s, 2005.
- [Derived] Fox E, Patel S, Wathen JK, Schuetze S, Chawla S, Harmon D, Reinke D, Chugh R, Benjamin RS, Helman LJ. Phase II study of sequential gemcitabine followed by docetaxel for recurrent Ewing sarcoma, osteosarcoma, or unresectable or locally recurrent chondrosarcoma: results of Sarcoma Alliance for Research Through Collaboration Study 003. Oncologist. 2012;17(3):321. doi: 10.1634/theoncologist.2010-0265. Epub 2012 Feb 23. PMID 22363068

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period began October 4, 2006 and was completed May 12, 2009. There were 11 SARC (Sarcoma Alliance for Research through Collaboration) sites participating. SARC sites are primarily academic institutions with Sarcoma programs.
Groups:
- Combination Chemotherapy: Gemcitibine 675 mg/m^2 given intravenous (IV) on day 1 and 8; docetaxel 75 mg/m^2 given IV on day 8 after gemcitibine. Each cycle is 21 days. Cycles of chemotherapy administered until off study criteria met.
Period: Overall Study
Arm/Group | Combination Chemotherapy
Started | 54
Completed | 53 (One patient in the chondrosarcoma subtype was not evaluable.)
Not Completed | 1
Not completed — not evaluable | 1

BASELINE CHARACTERISTICS:
Arm/Group | Combination Chemotherapy
Number analyzed (Participants) | 54
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 42
  >=65 years | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 43 (19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 54

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Patients will be evaluated up to 4 time points(after 2,4,8 and 12 cycles of therapy), each cycle is 21 days. Per RECIST 1.0 and assessed by CT/MRI disease status will be categorized as R=CR/PR(response), F=progressive disease or death(failure), or S(stable disease=neither R nor F) based on the change from baseline. A patient with outcome R or F at any stage is scored as having that overall outcome, a patient with outcome S is re-evaluated after subsequent cycles of therapy. Patients who receive more than 14 cycles of therapy will be scored as the outcome at completion of cycle 14.
Time Frame: After 2, 4, 8 and 12 cycles of therapy, each cycle is 21 days
Population: Analysis per protocol. One patient with chondrosarcoma was ineligible due to lack of measurable disease at enrollment.
Measure: Number; unit: participants
Groups:
- Ewing's Sarcoma; Osteosarcoma; Chondrosarcoma: Combination chemotherapy
Arm/Group | Ewing's Sarcoma | Osteosarcoma | Chondrosarcoma
Number analyzed (Participants) | 14 | 14 | 25
participants | 6 | 5 | 14

2. Secondary Outcome: Time to Progression
Description: Stable disease is measured from the start of the treatment until the criteria for disease progression are met, taking as reference the smallest measurements recorded since the treatment started. The clinical relevance of the duration of stable disease varies for different tumor types and grades. Bayesian statistical model is used. Timepoints for evaluation are post-cycle 2, 4, 8 and 12 using RECIST 1.0 criteria.
Time Frame: post-cycle 2, 4, 8 and 12
Population: Analysis not completed. One patient with chondrosarcoma was ineligible due to lack of measurable disease at enrollment.
Measure: Number; unit: months
Arm/Group | Ewing's Sarcoma | Osteosarcoma | Chondrosarcoma
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Toxicity as Assessed by NCI CTCAE v3.0
Description: Toxicity was graded according to Common Terminology Criteria for Adverse Events v.3.0 (CTCAE v.3.0). For gemcitabine or docetaxel related grade 3 or 4 non-hematological toxicities or hematological toxicities (grade 3 or 4 neutropenia for ≥ 7 days, grade 4 thrombocytopenia, or any platelet transfusion), both agents were withheld until the toxicity was ≤ grade 1. If the toxicity recovered to ≤ grade 1 by cycle day 35, the dose of both agents was reduced for all subsequent cycles. If the toxicity did not resolve by day 35, protocol therapy was discontinued.
Time Frame: Throughout the study
Population: Analysis per protocol. One patient with chondrosarcoma was ineligible due to lack of measurable disease at enrollment.
Measure: Number; unit: participants
Arm/Group | Ewing's Sarcoma | Osteosarcoma | Chondrosarcoma
Number analyzed (Participants) | 14 | 14 | 25
participants
  Toxicity | 4 | 3 | 5
  No Toxicity | 10 | 11 | 20

4. Secondary Outcome: Pharmacokinetics of Gemcitabine Alone and Gemcitabine Followed by Docetaxel at Protocol Specified Timeframe in Participants Enrolled on Study
Description: Blood samples for the determination of gemcitabine (and its metabolite dFdU) will be obtained prior to infusion, at 75 and 85 minutes (steady state), and 95 105 and 120 minutes, after the start of the 90 minute infusion on day 1 and day 8 of cycle 1. On day 8, docetaxel pharmacokinetics will be performed prior to infusion, 55 minutes (5 minutes prior to the end of infusion), 30 minutes post infusion, 5 hr and 24hr post infusion.
Time Frame: Gemcitibine: 0hr, 75, 85, 95, 105 and 120 min after the start of the 90 minute infusion; docetaxel: 0hr, 55 min, 30 min post infusion, 5hr and 24hr post infusion.
Population: There were insufficent samples obtained to analyze pharmacokinetics.
Measure: Number; unit: participants
Arm/Group | Ewing's Sarcoma | Osteosarcoma | Chondrosarcoma
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 years, 9 months
Arm/Group | Combination Chemotherapy
Serious Adverse Events (participants affected / at risk) | 12/53
Other Adverse Events (participants affected / at risk) | 36/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Chemotherapy (N=53)
cellulitis (Skin and subcutaneous tissue disorders) | 2 (3)
fever (Infections and infestations) | 3 (3)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 3 (3)
elevated WBC (Blood and lymphatic system disorders) | 1 (1)
pneumonia (Infections and infestations) | 3 (3)
hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
myositis (Musculoskeletal and connective tissue disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1)
confusion (Nervous system disorders) | 1 (1)
sepsis (Infections and infestations) | 1 (1)
pericardial effusion (Cardiac disorders) | 1 (1)
cardiac tamponade (Cardiac disorders) | 1 (1)
chest pain (Cardiac disorders) | 1 (1)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Combination Chemotherapy (N=53)
Grade 4 hematologic (Blood and lymphatic system disorders) | 14 (24)
Grade 3 hematologic (Blood and lymphatic system disorders) | 22 (58)

LIMITATIONS AND CAVEATS:
Since this design did not specify a rule for declaring the treatment as "active" a direct comparison to a standard 2 stage phase 2 design is not appropriate.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less